CLINICAL TRIAL: NCT05469113
Title: An Open-Label, Fixed-Sequence Study to Evaluate the Effect of Multiple Doses of LOXO-292 on the Single Dose Pharmacokinetics of Repaglinide in Healthy Adult Subjects
Brief Title: A Study of Effects of Selpercatinib (LY3527723) on Repaglinide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 17754; J2G-OX-JZJS (Other: Eli Lilly and Company); LOXO-RET-18026 (Other: Loxo Oncology, Inc.)
Record Dates: First submitted 2022-07-20; First posted 2022-07-21 (Actual); Results first posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Healthy
MeSH Terms: interventions — repaglinide; selpercatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1: Repaglinide (Experimental): * Day 1: Participants received single dose of 0.5 mg repaglinide tablet.
  Interventions: Drug: Repaglinide
- Period 2: Selpercatinib + Repaglinide (Experimental): * Day 1 to Day 9: Participants received 160 mg Selpercatinib capsule twice daily (BID).
  * Day 10: Participant received 160 mg Selpercatinib capsules BID co-administered with a single oral dose of 0.5 mg Repaglinide tablet on the morning of Day 10.
  Interventions: Drug: Repaglinide; Drug: Selpercatinib

INTERVENTIONS:
Drug: Repaglinide — Administered orally.
Drug: Selpercatinib — Administered orally.
  Other Names: LY3527723; LOXO-292
  Arms: Period 2: Selpercatinib + Repaglinide

SUMMARY:
The main purpose of this study is to assess the effect of selpercatinib on how fast repaglinide gets into the blood stream and how long it takes the body to remove it when administered in healthy participants. Information about safety and tolerability will be collected. The study will last up to 12 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kilograms per meter squared (kg/m²) and had a minimum weight of at least 50 kg at screening
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), and blood and urine laboratory test results that are acceptable for the study
* Hemoglobin (Hb) A1c value < 6.5 % at screening and fasting glucose ≤ 126 mg/dL.
* Males who are capable of fathering a child must agree to use one of the following methods of contraception from the time of the dose administration through 6 months after the last dose
* Female of non-childbearing potential only or must have undergone sterilization procedures at least 6months prior to the first dosing

Exclusion Criteria:

* History or presence of diabetes or history of prior episode(s) of hypoglycemia.
* Estimated creatinine clearance <90 mL/min at Screening or Check-in (Day -1, Period 1)
* Unable to refrain from or anticipates the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements for 14 days prior to the first dosing and through EOT or ET. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Period 1
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Started | 16 | 0
Safety Analysis Population (Received at Least One Dose of Study Drug) | 16 | 0
Completed | 16 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Started | 0 | 16 (Participants who completed Period 1, progressed to received treatment in Period 2.)
Safety Analysis Population (Received at Least One Dose of Study Drug) | 0 | 16 (2 participants discontinued the study on Day 3, and 1 participant discontinued study on Day 8 after receiving the Selpercatinib dose in Period 2. * Therefore, safety analysis population for Period 2: Selpercatinib + Repaglinide (Day 10) treatment includes only the remaining 13 participants.)
Completed | 0 | 13
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- All Participants: * Period 1: Participants received single dose of 0.5 mg Repaglinide tablet on Day 1.
  * Period 2: Participants received 160 mg Selpercatinib capsule twice daily (BID) from Day 1-10, and on Day 10 it was co-administered with a single oral dose of 0.5 mg Repaglinide tablet on the morning of Day 10.
Arm/Group | All Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Repaglinide
Time Frame: Period 1: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16 hours post dose); Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 16 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16 | 13
nanogram*hour per milliliter (ng*h/mL) | 9.409 (57.1) | 26.87 (53.2)

2. Primary Outcome: PK: Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-inf) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
nanogram*hour per milliliter (ng*h/mL) | 10.15 (51.3) | 27.31 (53.6)

3. Primary Outcome: PK: Percent of AUC0-inf Extrapolated (AUC%Extrap) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent AUC extrapolation
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
percent AUC extrapolation | 1.256 (43.8) | 1.258 (85.8)

4. Primary Outcome: PK: Maximum Observed Concentration (Cmax) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16 | 13
nanogram per milliliter (ng/mL) | 6.600 (77.4) | 12.11 (42.7)

5. Primary Outcome: PK: Time to Reach Maximum Observed Concentration (Tmax) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16 | 13
hours | 0.623 (47.3) | 0.854 (42.5)

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (Kel) of Repaglindide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: One per hour (1/h)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
One per hour (1/h) | 0.2406 (27.9) | 0.2036 (36.2)

7. Primary Outcome: PK: Apparent First-order Terminal Elimination Half-life (t½) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
hours | 2.881 (27.9) | 3.405 (36.2)

8. Primary Outcome: PK: Apparent Total Plasma Clearance After Oral (Extravascular) Administration (CL/F) of Repaglinide
Description: PK: CL/F of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hour (L/h)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
Liter per Hour (L/h) | 49.26 (51.3) | 18.31 (53.6)

9. Primary Outcome: PK: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of Repaglinide
Time Frame: as for outcome 1
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Period 1: Repaglinide | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 15 | 13
Liter (L) | 204.8 (53.6) | 89.92 (64.9)

10. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the 12 Hour (AUC0-12) of Selpercatinib
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16
ng*h/mL | 8424 (56.6)

11. Secondary Outcome: PK: Area Under the Concentration-time Curve, From Time 0 to the Last Observed Non-zero Concentration (AUC0-t) of Selpercatinib
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16
ng*h/mL | 8396 (56.7)

12. Secondary Outcome: PK: Maximum Observed Concentration (Cmax) of Selpercatinib
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16
ng/mL | 1476 (66.3)

13. Secondary Outcome: PK: Time to Reach Maximum Observed Concentration (Tmax) of Selpercatinib
Time Frame: Period 2: Day 1 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16
hours | 1.553 (25.9)

14. Secondary Outcome: PK: Area Under the Concentration-time Curve During a Dosing Interval (Tau) at Steady State (AUCtau) of Selpercatinib
Time Frame: Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 13
ng*h/mL | 33960 (45.0)

15. Secondary Outcome: PK: Maximum Observed Concentration at Steady-state (Cmax,ss) of Selpertcatinib
Time Frame: Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 13
ng/mL | 4082 (40.8)

16. Secondary Outcome: PK: Concentration Observed at the End of the Dosing Interval (Ctrough) of Selpercatinib
Time Frame: Period 2: Predose at Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome. 'Number analyzed' signifies participants with available data at specified timepoints.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 16
ng/mL
  Day 1 | 983.2 (225.43)
  Day 2 | 1509 (362.03)
  Day 3: number analyzed (Participants) | 14
  Day 3 | 1664 (529.60)
  Day 4: number analyzed (Participants) | 13
  Day 4 | 1842 (657.65)
  Day 5: number analyzed (Participants) | 14
  Day 5 | 1971 (642.36)
  Day 6: number analyzed (Participants) | 14
  Day 6 | 2039 (780.35)
  Day 7: number analyzed (Participants) | 14
  Day 7 | 2160 (771.22)
  Day 8: number analyzed (Participants) | 13
  Day 8 | 2034 (635.04)
  Day 9: number analyzed (Participants) | 13
  Day 9 | 2085 (762.09)

17. Secondary Outcome: PK: Time to Reach Maximum Observed Concentration at Steady-state (Tmax,ss) of Selpercatinib
Time Frame: Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 13
hours | 1.888 (29.6)

18. Secondary Outcome: PK: Apparent Total Plasma Clearance at Steady State After Oral/Extravascular Administration (CL,ss/F) of Selpercatinib
Time Frame: Period 2: Day 10 (Predose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 hours post dose)
Population: All participants who complied sufficiently with the protocol and displayed an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per Hours (L/h)
Arm/Group | Period 2: Selpercatinib + Repaglinide
Number analyzed (Participants) | 13
Liter per Hours (L/h) | 4.711 (45.0)

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to Day 2 for Period 1; up to Day 11 for Period 2)
Description: Safety analysis population: All participants who received at least one dose of study drug.
  * 2 participants discontinued the study on Day 3, and 1 participant discontinued study on Day 8 after receiving the Selpercatinib dose in Period 2. Therefore, safety analysis population for Period 2: Selpercatinib + Repaglinide (Day 10) treatment includes only the remaining 13 participants.
Groups:
- Period 1: Repaglinide (Day 1): * Day 1: Participants received single dose of 0.5 mg repaglinide tablet.
- Period 2: Selpercatinib (Day 1 to Day 9): * Day 1 to Day 9: Participants received 160 mg Selpercatinib capsule twice daily (BID).
- Period 2: Selpercatinib + Repaglinide (Day 10): * Day 10: Participant received 160 mg Selpercatinib capsules BID co-administered with a single oral dose of 0.5 mg Repaglinide tablet on the morning of Day 10.
Arm/Group | Period 1: Repaglinide (Day 1) | Period 2: Selpercatinib (Day 1 to Day 9) | Period 2: Selpercatinib + Repaglinide (Day 10)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 7/16 | 7/16 | 11/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Period 1: Repaglinide (Day 1) (N=16) | Period 2: Selpercatinib (Day 1 to Day 9) (N=16) | Period 2: Selpercatinib + Repaglinide (Day 10) (N=13)
Blood glucose decreased (Investigations) | 5 | 0 | 8
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 3
Fatigue (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT05469113/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05469113/SAP_001.pdf